CLINICAL TRIAL: NCT06384599
Title: Adagio Medical VT Cryoablation System Post-Market Clinical Follow-up (PMCF) Study
Brief Title: VT Cryoablation System Post-Market Clinical Follow-up (PMCF) Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adagio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-190
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Tachycardia
Keywords: Monomorphic Ventricular Tachycardia; VT; Cryoablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VT Cryoablation Arm (Experimental): all subjects will receive a cryoablation procedure with the VT System and be followed up for 6-month
  Interventions: Device: VT Cryoablation System

INTERVENTIONS:
Device: VT Cryoablation System — All subjects will receive a cryoablation procedure using the VT Cryoablation System (catheter, stylets, and console)

SUMMARY:
The PMCF is a prospective, single-arm, multi-center, controlled study of up to 130 patients designed to collect safety and performance data regarding the use of the Adagio VT Cryoablation System in the treatment of recurrent ventricular tachycardia.

DETAILED DESCRIPTION:
This VT Post-Market Clinical Follow-up (PMCF) study continues collecting additional information about the Adagio Medical VT Cryoablation System in real world clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* IC 1 Male or female the ages of ≥ 18 years
* IC 2 Planned ablation procedure according to the indication for use of the Adagio VT Cryoablation System
* IC 3 Subject willing to comply with study requirements and give informed consent
* IC4 Subject has or will be receiving an ICD prior to hospital discharge

Exclusion Criteria:

* EC 1 In the opinion of the investigator, any known contraindication to a ventricular tachycardia procedure with the Adagio VT Cyroablation System as indicated in the device Instructions For Use (IFU)
* EC 2 Subject is enrolled in a study that has not been approved for concurrent enrollment by the sponsor
* EC 3 Any other condition that, in the judgement of the investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, terminal illness with a life expectancy of less than six months, extensive travel away from the research center)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary Performance Endpoint | 6 months
  Freedom from ventricular tachycardia or appropriate ICD intervention until the end of the 6 month follow up period
Primary Safety Endpoint | 30 Days
  Freedom from device / procedure related major adverse events (MAE) during and after the ablation procedure through 30 days follow up. MAEs include:
  * Death
  * MI
  * Cardiac perforation / pericardial tamponade
  * Cerebral infarct or systemic embolism
  * Major bleeding requiring transfusion
  * Heart valve damage resulting in moderate to severe regurgitation
  * Access site complications requiring surgical intervention
  * Pericarditis
  * Heart block requiring a pacemaker implant
  * Other serious adverse device effects (SADEs).

SECONDARY OUTCOMES:
Secondary Performance Endpoint | During the procedure
  Analysis of the proportion of subjects with non-inducible clinical monomorphic VT at the conclusion of the initial cryotherapy ablation procedure.
Secondary Safety Endpoint | 6 months
  Freedom from serious adverse events at 6M following discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom